CLINICAL TRIAL: NCT07029165
Title: Neurovascular Control of Renal Blood Flow During Exercise in Older African American Adults
Brief Title: Kidney Blood Flow During Exercise in Older African American Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Rachel Drew, Associate Professor, University of Massachusetts, Boston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 3298; P20240000057554 (Other Grant/Funding Number: University of Massachusetts Boston)
Record Dates: First submitted 2025-06-04; First posted 2025-06-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Exercise; Cold stress; Mental stress
MeSH Terms: conditions — Motor Activity; Stress, Psychological | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- African American Adults (Experimental): African American adults will undergo the interventions of acute exercise, a cold pressor test, and a mental stress test while beat-to-beat renal blood flow velocity, mean arterial blood pressure, and heart rate are recorded.
  Interventions: Other: Acute exercise; Other: Cold pressor test; Other: Mental stress test
- White Adults (Experimental): White adults will undergo the interventions of acute exercise, a cold pressor test, and a mental stress test while beat-to-beat renal blood flow velocity, mean arterial blood pressure, and heart rate are recorded.
  Interventions: Other: Acute exercise; Other: Cold pressor test; Other: Mental stress test

INTERVENTIONS:
Other: Acute exercise — Participants will lie in a semi-supine position with their feet attached to the pedals of a custom-arranged cycle ergometer. Participants' 40% heart rate reserve will be calculated, giving the target value to achieve during exercise based on appropriate resistance applied on the cycle ergometer, corresponding to a moderate exercise intensity. After a 5-minute resting baseline, participants will perform dynamic cycling exercise at steady state for up to 20 minutes. They will then stop exercising, and there will be a 5-minute recovery period. Beat-to-beat renal blood flow velocity (Doppler ultrasound), mean arterial blood pressure (finger photoplethysmographic cuff), and heart rate (electrocardiogram) will be recorded throughout. A rating of perceived exertion will be taken from participants during the last 30 seconds of steady-state cycling exercise.
Other: Cold pressor test — Participants will lie in a semi-supine position, and after a 3-minute resting baseline, participants will have their hand immersed in ice water for 2 minutes. This cold pressor test represents the non-exercise, physical sympathetic stressor. Participants' hand will then be removed from the ice water, followed by a 3-minute recovery period. Beat-to-beat renal blood flow velocity (Doppler ultrasound), mean arterial blood pressure (finger photoplethysmographic cuff), and heart rate (electrocardiogram) will be recorded throughout. Ratings of hand pain and cold perception will be taken from participants during the last 30 seconds of the cold pressor test.
Other: Mental stress test — Participants will lie in a semi-supine position, and after a 3-minute resting baseline, participants will perform a mental arithmetic task for 5 minutes. This mental stress test represents the non-exercise, psychological sympathetic stressor. Participants will be instructed to subtract a given number from a randomly selected three-digit number and verbally state their answer and continue to do so for the duration of the test. Participants will be instructed to state their answers as quickly and accurately as possible. Participants will then stop the arithmetic task, and a 3-minute recovery period will follow. Beat-to-beat renal blood flow velocity (Doppler ultrasound), mean arterial blood pressure (finger photoplethysmographic cuff), and heart rate (electrocardiogram) will be recorded throughout. A rating of perceived stress will be taken from participants during the last 30 seconds of the mental stress test.

SUMMARY:
The goal of this preliminary study is to learn if healthy older African American (AA) adults have a larger change in their kidney blood flow during exercise compared to White (W) adults. The main questions that this study aims to answer are:

* Do healthy older AA adults have a larger decrease in kidney blood flow during exercise compared to W adults?
* Do healthy older AA adults have a larger decrease in kidney blood flow during other types of stress compared to W adults?

During one visit in the research lab, participants will:

* Perform cycling exercise while lying down
* Undergo a cold hand test
* Perform a mental math test

Completing this preliminary study will help researchers to understand more about why many AA adults have heart and kidney problems, so future research can study ways to reduce the number of AA adults who have these health issues.

DETAILED DESCRIPTION:
Racial disparities exist in the development of high blood pressure and heart and kidney disease. Over the last 25 years, African American (AA) adults have had the greatest prevalence of high blood pressure compared to any other racial identity group in the United States. In 2015, ~100,000 AA adults died from heart disease, accounting for one-third of all deaths in this population. AA adults also have a 2-3-times higher lifetime risk for developing end-stage kidney disease compared to White (W) adults. Further, advanced age is one of the most significant risk factors for developing high blood pressure, heart disease, and kidney disease. In 2013-2014, ~29% of deaths of adults aged 65 years or older were caused by heart disease, the leading cause of death in this population.

Elevated sympathetic nervous system activity is associated with increased incidence of heart and kidney disease. Physical activity, such as exercise, acutely increases sympathetic nervous system activity, notably directed towards the kidneys, resulting in reflex narrowing of small blood vessels inside the kidneys. This response reduces blood flow to the kidneys to deliver greater blood flow to the active skeletal muscles. Most of the research studies in this area have involved participant groups who were wholly or predominantly of W racial identity, with smaller proportions of individuals of other racial identities. This underrepresentation of non-W participants, including AA adults, has occurred despite the known health disparities such as the greater incidence of high blood pressure and heart disease and kidney disease experienced by these populations.

A larger decrease in kidney blood flow during exercise has been observed in patients with heart failure and peripheral arterial disease compared to healthy adults. However, it is not known whether the decrease in kidney blood flow during exercise is larger in healthy older AA adults compared to other racial identity groups. Given the greater level of chronic psychological stress often experienced by AA adults due to systemic racism and social and environmental factors, the associated cumulative negative impact on cardiovascular health could underlie a physiological difference observed between AA and W adults. Therefore, it is hypothesized that healthy older AA adults will exhibit a larger decrease in kidney blood flow during exercise compared to W adults. This greater response in older AA adults could be a significant factor contributing to the higher rates of heart and kidney disease in this population given the negative effect that this larger response could have over time, highlighting the clinical significance of this area.

The goal of this project is to collect preliminary data regarding the kidney blood flow response to exercise in healthy older AA compared to W adults. This will be achieved through the innovative use of Doppler ultrasound to noninvasively measure kidney blood flow in real time during cycling exercise in 6 healthy older AA adults and 6 healthy older W adults. The preliminary data collected in this project will be used to strengthen future proposals to secure external funding to complete this project on a larger scale. Findings from a larger-scale project will have important implications for developing preventative strategies to reduce the elevated risk of developing heart and kidney disease in the AA population.

ELIGIBILITY:
Inclusion Criteria:

* Self-report as either African American or White racial identity
* Born in United States
* Both biological parents identify as same racial identity as participant
* Recreationally active (participating in physical activity for at least 20 minutes per day, at least three times per week, but not training for competitive events)
* Fluent in English

Exclusion Criteria:

* Hispanic or Latino
* Females who are pregnant or lactating
* Cardiovascular or renal disease
* Hypertension (blood pressure of more than or equal to 130/80 mmHg)
* Diabetes
* Obesity (body mass index of more than or equal to 30 kg/m2)
* Smoker/Tobacco user
* Acute medical conditions
* Taking prescribed cardiovascular, antihypertensive, or renal medications

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female
Enrollment: 12 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in renal vascular resistance during acute exercise | Pre-acute exercise and during 5 minutes of steady-state exercise
  For the acute exercise intervention, the percent change from pre-acute exercise to during steady-state exercise will be assessed.
Change in renal vascular resistance during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the percent change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in renal vascular resistance during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the percent change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.

SECONDARY OUTCOMES:
Change in renal blood flow velocity during acute exercise | Pre-acute exercise and during 5 minutes of steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in mean arterial blood pressure during acute exercise | Pre-acute exercise and during 5 minutes of steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in systolic blood pressure during acute exercise | Pre-acute exercise and during 5 minutes of steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in diastolic blood pressure during acute exercise | Pre-acute exercise and during 5 minutes of steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in heart rate during acute exercise | Pre-acute exercise and during 5 minutes of steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in cardiac output during acute exercise | Pre-acute exercise and during 5 minutes of steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in stroke volume during acute exercise | Pre-acute exercise and during 5 minutes of steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in total peripheral resistance during acute exercise | Pre-acute exercise and during 5 minutes of steady-state exercise
  For the acute exercise intervention, the absolute change from pre-acute exercise to during steady-state exercise will be assessed.
Change in renal blood flow velocity during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in mean arterial blood pressure during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in systolic blood pressure during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in diastolic blood pressure during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in heart rate during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in cardiac output during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in stroke volume during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in total peripheral resistance during cold pressor test | Pre-cold pressor test to after 30, 60, 90, and 120 seconds of cold pressor test
  For the cold pressor test intervention, the absolute change from pre-cold pressor test to 30-second intervals during the cold pressor test will be assessed.
Change in renal blood flow velocity during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in mean arterial blood pressure during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in systolic blood pressure during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in diastolic blood pressure during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in heart rate during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in cardiac output during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in stroke volume during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.
Change in total peripheral resistance during mental stress test | Pre-mental stress test to after 1, 2, 3, 4, and 5 minutes of mental stress test
  For the mental stress test intervention, the absolute change from pre-mental stress test to 1-minute intervals during the mental stress test will be assessed.

OTHER OUTCOMES:
Rating of perceived exertion during acute exercise | During last 30 seconds of steady-state exercise
  For the acute exercise intervention, the rating will be taken during the last 30 seconds of steady-state exercise. The Borg Scale of Perceived Exertion will be used, with which a rating from 6 to 20 will be taken, with 6 representing no exertion and 20 representing maximal exertion.
Rating of hand pain during cold pressor test | During last 30 seconds of cold pressor test
  For the cold pressor test intervention, the rating will be taken during the last 30 seconds of the cold pressor test. A scale from 0 to 10 will be used to take the rating, with 0 representing no pain and 10 representing the worst possible pain.
Rating of cold perception during cold pressor test | During last 30 seconds of cold pressor test
  For the cold pressor test intervention, the rating will be taken during the last 30 seconds of the cold pressor test. A scale from 0 to -11 will be used to take the rating, with 0 representing no perceived cold and -11 representing unbearable cold.
Rating of perceived stress during mental stress test | During last 30 seconds of mental stress test
  For the mental stress test intervention, the rating will be taken during the last 30 seconds of the mental stress test. A scale from 0 to 4 will be used to take the rating, with 0 representing no perceived stress and 4 representing extremely stressful.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel C Drew, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (1):
- University of Massachusetts Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No